CLINICAL TRIAL: NCT02156427
Title: A Multicenter Double-blind Placebo-controlled Trial of Non-cultured Epidermal Cellular Grafting Versus Hyaluronic Acid for Repigmenting Stable Leukoderma (Vitiligo and Piebaldism)
Brief Title: Evaluation of Non-cultured Epidermal Cellular Grafting vs Hyaluronic Acid for Repigmenting Vitiligo and Piebaldism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13INT/VIT01
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Vitiligo; Piebaldism
MeSH Terms: conditions — Vitiligo; Piebaldism

STUDY DESIGN:
Intervention Model Description: double-blind, prospective, multicenter, randomised, controlled trial patient is his own control
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VITICELL (Experimental): In this arm, lesions will be treated by autologous epidermal cells suspension (containing hyaluronic acid) obtained after VITICELL kit's use, a class III medical device.
  Interventions: Device: VITICELL
- PLACEBO (Placebo Comparator): In this arm, lesions will be treated by a suspension of hyaluronic acid without epidermal cells.
  Interventions: Device: PLACEBO

INTERVENTIONS:
Device: VITICELL — graft of autologus cells (kaeratonicytes and melanocytes) obtained after trypsinization of thin skin biopsy resuspended into hyaluronic acid
  Arms: VITICELL
Device: PLACEBO — hyaluronic acid alone
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to assess the efficacy of autologous epidermal cells suspension grafting using a newly developed device named VITICELL® compared to placebo.

The secondary objective is to evaluate safety of VITICELL® and global satisfaction of patient and investigator.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years old with a diagnosis of non-scaring leukoderma that has been stable over the last 2 years (non-segmental, segmental vitiligo and piebaldism)
* For non-segmental vitiligo: symmetrical vitiligo lesions, or parts of a lesion. A part of at least 1 cm2 (1 x 1 cm), but preferable 4 cm2 (2x2 cm) and preferably in the center of each lesions (left/right) should be treated.

The minimum distance between the normal pigmented skin and the test area should preferably be at least 0.5 cm.

* For segmental vitiligo lesion and piebaldism: all lesions possible if two parts of at least 1 cm2 (1 x 1 cm), but preferably 4 cm2 (2 x 2 cm) in the lesion can be treated. The minimum distance between the 2 areas should be 2 cm and between test areas and to the normal pigmented skin preferably at least 0.5 cm.
* Medical treatments of vitiligo failed (in case of vitiligo: at least cream treatment for 6 months).
* Absence of infected lesion
* Negative serology (HIV-hepatitis B and C- Syphilis)
* Without treatment one month for cream and 3 months for phototherapy

Exclusion Criteria:

* Hypersensibility to local anaesthetics or one of the components of the device (trypsin, hyaluronic acid)
* Indication against biopsies
* Patient with a history of melanoma
* Positive serology (ongoing serious systemic disease, herpes, HIV, hepatitis B and C-Syphilis)
* Positive pregnancy test
* History of keloidal scars and presence of Koebner's phenomenon (type 1 and type 2b)
* Infected lesion
* Test areas not on fingers and toes vitiligo areas in case of non-segmental vitiligo
* Test areas not on facial non segmental vitiligo
* Pregnant women, or lactating
* Age <18years
* Major deprived of their freedom by administrative or legal decision, or being the subject of a legal protection measure, or out of state to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Rate of successful repigmentation | at month 6
  succesful repigementation define as more than or equal to 50% repigmentation of the treated area

SECONDARY OUTCOMES:
Rate of successful repigmentation | at month 12
  succesful repigementation define as more than or equal to 50% repigmentation of the treated area

OTHER OUTCOMES:
Number of adverse events in each group | Day 0/Day 6-7/Month 3/6/9/12
Mean reduction of treated area | Month 3/6/9/12
  calculated in pourcentage from baseline
Variation of area size | Day 0/Month 3/6/9/12
  Size in cm² measured at each visit
Patient and physician satisfaction | Month12
  Likert scale ranging from 1 to 5 (1=Not at all satisfied / 2=Slightly satisfied / 3=Moderately satisfied / 4=Very satisfied / 5=Extremely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Nanja Van Geel, Pr, Principal Investigator — Gent hospital
Locations (5):
- Department of Dermatology - Ghent University Hospital, Ghent, Belgium
- France (3):
  - University Hospital Center of Bordeaux, Bordeaux
  - CHU Le Mans, Le Mans
  - Dr Michel PASCAL, Paris
- San Gallicano Dermatological Institute, Roma, Italy